CLINICAL TRIAL: NCT03549052
Title: Right Ventricular Function After Mitral Valve Replacement in Rheumatic Heart Disease Patients With Pulmonary Hypertension: Short Term Follow up
Brief Title: Right Ventricular Echo Assessment in Mitral Valve Replacement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed M. Nasr, Assistant Lecturer Cardiothoracic surgery, Assiut University
Other Study IDs: Echo in mitral valve diseases
Record Dates: First submitted 2018-05-22; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Right Ventricular Dysfunction; Rheumatic Heart Disease
MeSH Terms: conditions — Ventricular Dysfunction, Right; Rheumatic Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rheumatic heart disease remains a major health problem in developing countries. It is the most important sequel of rheumatic fever and occurs in about 30% of patients with rheumatic fever.Rheumatic heart disease presents with different degrees of pancarditis and associated valve failure. Involvement of the mitral leaflets can cause mitral regurgitation (MR) or stenosis and eventually can lead to heart failure. Mitral repair or replacement is therefore recommended before left ventricular (LV) dysfunction develops.

Study Objectives/Specific Aims Overall Goal: To determine the benefit the patient with pulmonary hypertension will get from mitral valve replacement as regard function improvement and remodeling of the right ventricle.

* Objective1: Identify risk factors that are predictive of outcomes.(Type and severity of Mitral valve pathology , severity of pulmonary hypertension, tricuspid regurge, preoperative RV dysfunction)
* Objective2: Determine the value of management strategies (Mitral valve replacement in pulmonary hypertension i.e. : decrease RV pressure overload and enhance RV remodeling)
* Objective3: Assessment of the outcomes clinically & Echocardiographically : postoperative results during hospital stay and follow up (short term up to 3 months).

DETAILED DESCRIPTION:
In 1994, it was estimated that 12 million individuals had RF and RHD worldwide , and at least 3 million had congestive heart failure (CHF) that required repeated hospital admissions. A large section of the individuals with CHF required cardiac valve surgery within 5-10 years . The mortality rate for RHD varied from 0.5 per 100 000 population in Denmark, to 8.2 per 100 000 population in China , and the estimated annual number of deaths from RHD for 2000 was 332000 worldwide . The mortality rate per 100 000 population varied from 1.8 in the WHO Region of the Americas, to 7.6 in WHO South-East Asia Region. The disability-adjusted life years (DALYs)1 lost to RHD ranged from 27.4 DALYs per 100 000 population in the WHO Region of the Americas, to 173.4 per 100 000 population in the WHO South-East Asia Region. An estimated 6.6 million DALYs are lost per year worldwide.

THE PATHOLOGY OF RHEUMATIC MITRAL VALVE DISEASE Rheumatic mitral valves shows a different set of lesions by comparison with degenerative valves, because of the characteristic inflammatory process, which results in thickening of the leaflets and other components of the mitral valve apparatus, of variable degrees, and distorts and impairs the movements of the valve. So, the disease appears here in two forms - stenosis and regurgitation, or a combination of both.

In the case of valve regurge, the most frequent lesion is prolapse of the anterior leaflet, which is present in more than 90% of young patients and is most often caused by elongated chordae to its central and medial areas (A2 and A3). In contrast to degenerative disease, posterior leaflet prolapse is practically not found, except in cases with ruptured chordae due to infective endocarditis. On the contrary, this leaflet is often shortened in its width, sometimes resumed to a very narrow and thick strip of tissue. In more complicated cases, the chordae may be thick and retracted, as may also be the papillary muscles, and the commissures may be fused in varying degrees. Often, the leaflets and subvalvular apparatus are a continuous mass of fibrous tissue. Lastly, the annulus is dilated in 95% of the patients. It is widely accepted that dilatation occurs essentially in the posterior segment of the annulus, although there is some evidence that it may also occur in the anterior segment, especially in dilated cardiomyopathy.

Pulmonary hypertension and valvular heart disease Valvular Heart Disease VHD is a common etiology of pulmonary hypertension, which may result from many mechanisms as an increase in pulmonary vascular resistance, pulmonary blood flow, or pulmonary venous pressure. The chronic rise in pulmonary arterial pressure (PAP) often leads to right ventricular (RV) pressure overload and subsequent RV failure. When present, PH is a marker of poor outcome in VHD. Assessment of the presence and severity of Pulmonary hypertension thus has an important role in the risk stratification and therapeutic management of VHD.

The sure diagnosis of PH related to VHD is based on the following criteria: mean PAP 25 mm Hg together with an abnormally high pulmonary capillary wedge pressure (PCWP) >15 mm Hg or left ventricular (LV) end-diastolic pressure >18 mm Hg in the context of significant VHD. When pulmonary venous congestion is the main determinant of PH, PH is named isolated post-capillary PH or pulmonary venous hypertension.

PATHOPHYSIOLOGY Increase in LV filling pressure and left atrial (LA) pressure leads to a passive rise in backward pressure of the pulmonary vein. Persistently elevated pulmonary venous pressure can favor fragmentation of the structure and result in "alveolar capillary stress failure," accompanied by capillary leakage and acute alveolar edema. This acute phase is reversible, but long-term persistence of high pulmonary venous pressure may provocate some degree of irreversible remodeling of the alveolar capillary membrane, with excessive deposition of type IV collagen. Plus, chronic elevated pulmonary venous pressure progressively and passively increases PAP and concomitantly produces pathological changes in pulmonary veins. and arteries, leading to increased pulmonary vascular resistance . The pathophysiology of PH in VHD thus involves progressive structural alteration of the pulmonary vascular bed mediated by the potent vasoconstrictor endothelin-1 . An increase in pulmonary-arterial vasoconstriction and systolic PAP results into RV dilation and hypertrophy. The RV failure is associated with tricuspid annulus dilation and an increase in tricuspid regurgitation severity, which further acerbates RV dysfunction. At the decompensated phase, systolic PAP can decrease despite the increase in pulmonary vascular resistance, due to the fall in RV stroke volume related to advanced RV failure.

After treatment, the reversibility of PH depends on the type, severity, and chronicity of VHD, as well as the underlying pathophysiological adaptations. For instance, in mitral stenosis (MS), a rapid decrease in PAP is observed after relief of the stenosis, whereas a longer time could be required in other VHDs, especially when PH is linked to volume overload, as in mitral regurgitation (MR). Right ventricular function assessment The right ventricle has long been neglected, yet it is RV function that is strongly associated with clinical outcomes in many conditions. Although the left ventricle has been studied extensively, with established normal values for dimensions, volumes, mass, and function, measures of RV size and function are lacking. The relatively predictable left ventricular (LV) shape and standardized imaging planes have helped establish norms in LV assessment. There are, however, limited data regarding the normal dimensions of the right ventricle, in part because of its complex shape. The right ventricle is composed of 3 distinct portions: the smooth muscular inflow (body), the outflow region, and the trabecular apical region. Volumetric quantification of RV function is challenging because of the many assumptions required. As a result, many physicians rely on visual estimation to assess RV size and function.

The basics of RV dimensions and function were included as part of the ASE and European Association of Echocardiography recommendations for chamber quantification published in 2005. This document, however, focused on the left heart, with only a small section covering the right-sided chambers. Since this publication, there have been significant advances in the echocardiographic assessment of the right heart. In addition, there is a need for greater dissemination of details regarding the standardization of the RV echocardiographic examination .

PERIOPERATIVE ASSESSMENT OF THE RV In cardiac surgery, right heart catheterization and echocardiography play an essential and complementary role in the assessment of RV structure and function. Both provide useful information that may help tailor the anesthetic and surgical approach and provide guidance in the management of hemodynamically unstable patients. Hemodynamically, Right ventricular dysfunction or failure is usually recognized in the presence of a right atrial pressure (RAP) _8-10 mm Hg or a RAP to pulmonary capillary wedge pressure _0.8 (isolated RV failure) and/or a low cardiac index (_2.2 L _ min_1 _ m_2). Increasing RAP may also be a sign of impeding RV failure. echocardiography also provides useful information on RV and pulmonary structure, valvular function and pericardial physiology.

The echocardiographic evaluation of the RV is more challenging than that of the left ventricle. The main difficulties encountered may be explained by 1) the complex shape of the RV, 2) heavy apical trabeculations of the RV, which limits endocardial surface recognition, and 3) the marked load dependence of several indices of RV function. Despite these limitations, a comprehensive assessment of the RV may provide important data into its contractility, preload, and afterload.

Lastly and as recommended by the American society of Echocardiography Endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography in 2010 guidelines all studies, the sonographer and physician should examine the right heart using multiple acoustic windows, and the report should represent an assessment based on qualitative and quantitative parameters. The parameters to be performed and reported should include a measure of right ventricular (RV) size, right atrial (RA) size, RV systolic function (at least one of the following: fractional area change [FAC], S', and tricuspid annular plane systolic excursion [TAPSE]; with or without RV index of myocardial performance [RIMP]), and systolic pulmonary artery (PA) pressure (SPAP) with estimate of RA pressure on the basis of inferior vena cava (IVC) size and collapse.

So in this study we will focus on right ventricular function and performance after performing Mitral valve replacement to the rheumatic heart disease patients associated with pulmonary hypertension either mild or severe, to put a hand on the extent of benefit the patient who developed pulmonary hypertension will get from mitral valve replacement as regard function improvement and remodeling of the right ventricle and the proper timing of surgery.

ELIGIBILITY:
Inclusion Criteria:

* All ages will be accepted.
* Isolated mitral valve lesion either stenosis or regurge.
* Good LV function (EF <45%).
* Any degree of tricuspid valve regurge..

Exclusion Criteria:

* Concomitant Aortic valve lesion needs replacement.
* Poor LV function (Low EF> 45%).
* Other causes of pulmonary hypertension i.e.: (Chronic obstructive or restrictive pulmonary disease, connective tissue disease and chronic thromboembolism).
* Emergency and Redo operations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who presented to our department of Cardiothoracic surgery, Assiut University hospitals from May 2018 to April 2020 and who are candidate for mitral valve replacement and meet the listed inclusion and exclusion criteria will be eligible for the study. The charts will be reviewed and eligible patients will be filtered. The needed variables will be entered into our data base, for later data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between echocardiographic parameters of the RV, measured with TTE , preoperative and short term post operative | Baseline-1 Week-3 months
  change in TAPSE (Tricuspid annular plane systolic excursion )

SECONDARY OUTCOMES:
postoperative Response in right ventricular function parameter S' Change in S' | Baseline-1 Week-3 months
  TDI (Tissue doppler imaging) across the lateral tricuspid annulus : peaked S' velocity
Postoperative Response in right ventricular function parameter RVFAC | Baseline-1 Week-3 months
  change in RVFAC : Right ventricular calculated ejection fraction by mean of change in RV systolic and diastolic volumes
Postoperative Response in right ventricular function parameter pulmonary artery systolic pressure | Baseline-1 Week-3 months
  PASP measured by CW doppler across tricusped valve regurgetant jet
Postoperative right atrial pressure assesment | Baseline-1 Week-3 months
  RA diamter and IVC collapsability in cm
Evaluation of reverse right ventricle (RV) remodelling | Baseline-1 Week-3 months
  The evaluation of reverse right ventricle (RV) remodelling, assessed as reduction/modification of the end diastolic and end systolic RV diameters with respect to pre-surgery
Residual TR | Baseline-1 Week-3 months
  Percentage of patients with moderate to severe TR at 3 months after surgery

OTHER OUTCOMES:
NYHA Class | 3 months
  Modification of NYHA class at 3 months after surgery
Mortality | up to 3 months of intervention
  Mortality within hospital stay or 3 months postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. EL_Minshawy, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Naeije R. Assessment of right ventricular function in pulmonary hypertension. Curr Hypertens Rep. 2015 May;17(5):35. doi: 10.1007/s11906-015-0546-0. PMID 25833458
- [Result] Kjaergaard J. Assessment of right ventricular systolic function by tissue Doppler echocardiography. Dan Med J. 2012 Mar;59(3):B4409. PMID 22381093
- [Result] Ling LF, Marwick TH. Echocardiographic assessment of right ventricular function: how to account for tricuspid regurgitation and pulmonary hypertension. JACC Cardiovasc Imaging. 2012 Jul;5(7):747-53. doi: 10.1016/j.jcmg.2011.08.026. No abstract available. PMID 22789943
- [Result] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Result] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: II. Pathophysiology, clinical importance, and management. Anesth Analg. 2009 Feb;108(2):422-33. doi: 10.1213/ane.0b013e31818d8b92. PMID 19151265
- [Result] Magne J, Pibarot P, Sengupta PP, Donal E, Rosenhek R, Lancellotti P. Pulmonary hypertension in valvular disease: a comprehensive review on pathophysiology to therapy from the HAVEC Group. JACC Cardiovasc Imaging. 2015 Jan;8(1):83-99. doi: 10.1016/j.jcmg.2014.12.003. PMID 25592699
- [Result] Bayat F, Aghdaii N, Farivar F, Bayat A, Valeshabad AK. Early hemodynamic changes after mitral valve replacement in patients with severe and mild pulmonary artery hypertension. Ann Thorac Cardiovasc Surg. 2013;19(3):201-6. doi: 10.5761/atcs.oa.11.01865. Epub 2012 Oct 15. PMID 23064658
- [Result] Kret M, Arora R. Pathophysiological basis of right ventricular remodeling. J Cardiovasc Pharmacol Ther. 2007 Mar;12(1):5-14. doi: 10.1177/1074248406298293. PMID 17495253